CLINICAL TRIAL: NCT01441531
Title: Efficacy of Gabapentin in Prevention of Tourniquet Pain and Hypertension During Orif of Tibia Fracture Under General Anesthesia
Brief Title: Efficacy of Gabapentin in Prevention of Tourniquet Pain and Hypertension
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to recruit patient due to surgical case type. Not worth continuing study.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-28860
Record Dates: First submitted 2011-09-21; First posted 2011-09-27 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Tourniquet-induced Pain; Tourniquet-induced Hypertension
Keywords: narcotic use; Other Acute Pain
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin 600 mg po given 1 hour before surgery
  Interventions: Drug: gabapentin 600 mg po
- Placebo sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo pill given one hour before surgery

INTERVENTIONS:
Drug: gabapentin 600 mg po — Given one hour before surgery
  Arms: Gabapentin
Drug: Placebo pill given one hour before surgery — Placebo pill given
  Arms: Placebo sugar pill

SUMMARY:
The purpose of the study is to find out if taking a dose of gabapentin 600 mg by mouth (po) before surgery will help prevent the development of tourniquet pain and hypertension while the tourniquet is inflated during orif of tibia fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages 18-64
* ASA physical status 1-3
* Schedule for orif tibia fracture with use of pneumatic tourniquet

Exclusion Criteria:

* Allergy to study medications
* polytrauma
* lower extremity crush injury
* chronic opioid use
* sickle cell disease or trait
* peripheral vascular disease
* poorly controlled hypertension
* history of DVT/PE
* morbid obesity (BMI > 35)
* patient or surgeon refusal
* patient inability to properly describe postoperative pain to investigators

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of tourniquet-induced hypertension | During the tourniquet inflation time period
  Primary outcome is incidence of tourniquet-induced hypertension, which is defined as an increase of systolic or diastolic blood pressure > 30% from baseline. This will be looked at during the time of tourniquet inflation (from inflation to deflation) during the actual surgical procedure. Usual maximum inflation time is 120 minutes.

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  Postoperative pain scores for 24 hours after surgery
Narcotic use | 24 hours
  Total use of morphine, vicodin during 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ortiz, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States